CLINICAL TRIAL: NCT06704685
Title: A Randomized Controlled Trial on the Efficacy and Safety of Butylphthalide in Reducing Myocardial Infarction Size and Improving Outcomes in STEMI Patients After Primary PCI - A Prospective, Multicenter, Randomized, Placebo, Double-blinded End Trial.
Brief Title: A Randomized Controlled Trial on the Efficacy and Safety of Butylphthalide in Reducing Myocardial Infarction Size and Improving Outcomes in STEMI Patients After Primary PCI
Acronym: RISE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: CSPC Pharmaceutical Group Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202409176
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — 3-n-butylphthalide

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly assigned in a 1:1 ratio to two groups: a butylphthalide group and a placebo group.The Butylphthalide group received 100ml of butylphthalide injection twice a day for 7±2 days, followed by butylphthalide soft capsules (2 capsules, three times a day) from the day of discharge to day 30±2. The placebo group received the same dosage of butylphthalide injection and soft capsules placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide group (Experimental): The Butylphthalide group received 100ml of butylphthalide injection twice a day for 7±2 days, followed by butylphthalide soft capsules (2 capsules, three times a day) from the day of discharge to day 30±2.
  Interventions: Drug: Butylphthalide
- Placebo group (Placebo Comparator): The placebo group received 100ml of butylphthalide placebo injection twice a day for 7±2 days, followed by butylphthalide placebo soft capsules (2 capsules, three times a day) from the day of discharge to day 30±2.
  Interventions: Drug: Butylphthalide placebo

INTERVENTIONS:
Drug: Butylphthalide — Subjects who were initially diagnosed with STEMI and scheduled for PCI were randomly assigned to one of two groups in a 1:1 ratio: a butylphthalide group and a placebo group.
  Arms: Butylphthalide group
Drug: Butylphthalide placebo — Butylphthalide placebo
  Arms: Placebo group

SUMMARY:
This study is a prospective, randomized, placebo-double-blind, multicenter clinical trial. The purpose of this study is to investigate whether "butylphthalide +PCI" combined treatment mode on the basis of traditional drug therapy could reduce myocardial infarct size, improve cardiac function and long-term prognosis of patients with acute myocardial infarction, and verify the drug safety of butylphthalide in the treatment of STEMI within the window period of 12 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-75 years, encompassing both genders;
2. Patients presenting with an initial clinical diagnosis of acute ST-segment elevation myocardial infarction (STEMI), within a maximum time frame of 12 hours from the onset of pain to consideration for trial inclusion, who fulfill the criteria for percutaneous coronary intervention (PCI) and express their intention to undergo PCI;
3. The subject and their legal representative possess the capacity and willingness to provide informed consent by signing.

Exclusion Criteria:

1. Uncontrolled hypertension (systolic blood pressure≥200mmHg and/or diastolic blood pressure≥110mmHg);
2. Previous PCI or CABG;
3. Long-term use of loading doses of anticoagulant or antiplatelet drugs;
4. History of hemorrhagic stroke or ischemic stroke within 6 months, peptic ulcer, prolonged cardiopulmonary resuscitation (more than 10 minutes) within the last 6 weeks, surgery, or major trauma;
5. Known allergy to butylphthalide or excipients;
6. Patients with any of the following conditions: cardiogenic shock, chronic congestive heart failure NYHA class ≥III, severe hypotension, pulmonary insufficiency, severe hepatic and renal insufficiency;
7. History of congenital or acquired hemorrhagic diseases, coagulation factor deficiency diseases, thrombocytopenic diseases, etc. Or any of the following laboratory tests (INR > 2.0, platelet count < 100×109/L, Hb < 10g/dl);
8. Pregnancy, lactation, and planning to become pregnant within 30 days;
9. Severe mental disorder, alcohol dependence or inability to cooperate with informed consent and follow-up due to dementia;
10. Concurrent malignant tumor or severe systemic disease with expected survival time less than 30 days;
11. Have participated in or are currently participating in another clinical intervention study within 30 days before randomization;
12. Other reasons for not being eligible for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy in reducing myocardial infarct size in subjects with STEMI after primary PCI | 30±2 days post-randomization
  To evaluate the efficacy of butylphthalide injection versus placebo in reducing myocardial infarct size at day 30 in patients with STEMI after primary PCI.

SECONDARY OUTCOMES:
The proportion of no-reflow and severe slow flow events | 30±2 days post-randomization
  The proportion of no-reflow and severe slow flow events on day 30±2 after randomization (TFG<2 is defined as slow flow events and angiographic score).
The changes of ST-segment resolution in electrocardiogram | 7±2 days and 30±2 days post-randomization
  ST-segment resolution of electrocardiogram at 7±2 days and 30±2 days after randomization.
CMR imaging cardiac function indexes and cardiac color Doppler ultrasound related indexes | 30±2 days post-randomization
  CMR examination of microcirculation obstruction area, delayed enhancement phenomenon, left ventricular ejection fraction (LVEF%) and other CMR imaging cardiac function indicators and cardiac color Doppler ultrasound related indicators.
The decline of myocardial enzyme indexes | 7±2 days and 30±2 days post-randomization
  Myocardial enzyme indexes (CK-MB, troponin I or T) decline at 7±2 days and 30±2 days of randomization.
Proportion of combined vascular events | 30±2 days post-randomization
  Rate of combined vascular events (symptomatic stroke, recurrent myocardial infarction, vascular death) at 30±2 days after randomization.